CLINICAL TRIAL: NCT06354764
Title: Propensity to Hospitalize Patients From the ED in European Centers.An Observational Retrospective Quality-of-care Study
Brief Title: Propensity to Hospitalize Patients From the ED in European Centers.
Acronym: eCREAM-UC1
Status: Not yet recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Astir S.r.l. (Unknown); Centre Hospitalier Universitaire Vaudois (Other); Orobix Life S.r.l. (Unknown); Fondazione Bruno Kessler (Other)
Responsible Party: Sponsor
Other Study IDs: 8780-UC1
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Emergency Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults who attended the emergency department
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The peer-to-peer comparison means center-to-center comparison, which requires adjusting for possible differences among centers to be fair and convincing. The first step to reach this goal is to develop a predictive model that accurately estimates each patient's probability of being admitted, starting from clinical conditions and boundary variables. Such a model would make it possible to calculate, for each ED, the expected hospitalization rate; that is, the hospitalization rate that would have been observed if the ED had behaved like the average of the EDs that provided the data to build the model itself. Comparing the observed hospitalization rate in the single ED with the expected rate derived from the model provides a rigorous method of comparing the department with the average performance, taking into account the characteristics of the patients treated and the conditions under which the ED operated. In other words, the predictive model represents the benchmark against which each ED is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Arrived at emergency department between 1 January 2021 and 31 December 2023

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who arrived at participating emergency departments between January 1, 2021 and December 31, 2023
Sampling Method: Probability Sample
Enrollment: 162000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Create two separate databases | September 2024 - September 2025
  To create two separate databases (one for each of the two subgroups considered) on all patients who presenteding to the participating EDs over a defined period, containing the information considered important to study both the propensity to hospitalize these patients and their 30-day mortality
Multivariable models | September 2025 - September 2026
  To develop two multivariable models that predict the probability that patients presenting to the ED with dyspnea (first model) or after a TLoC (second model) will be admitted to the hospital
Adjusted comparison | September 2025 - September 2026
  To provide the participating EDs with an adjusted comparison of the hospitalization rates for the patients with selected symptoms, to improve the quality of care.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Bertolini, MD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri

IPD SHARING:
Plan to Share IPD: Yes
eCREAM-UCI1 will join the MIP (Medical Informatics Platform), developed in the Human Brain Project (HBP), to federate clinical data. The MIP is an open-source, GDPR-compliant, privacy-aware platform, enabling remote and federated analyses from datasets physically distributed in various hospitals, research centers, and biobanks, without moving the data outside their original storage site to a central repository. Patient identification data will be deleted from the databases before these are uploaded to the MIP platform, and no pseudo-identifier will be available.
  See https://mip.ebrains.eu/ for more details on the MIP.
Supporting Information: Study Protocol